CLINICAL TRIAL: NCT03115606
Title: Comparison of C-Mac D Blade and Fastrach Laryngeal Mask Airway on Cervical Spine Motion Conditions in Cervical Discectomy
Brief Title: Comparison of C-Mac D Blade and Fastrach Laryngeal Mask Airway on Cervical Spine Motion Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Associated professor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Diskapi3
Record Dates: First submitted 2017-03-26; First posted 2017-04-14 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Intubation Complication; Cervical Discopathy
Keywords: videolaryngoscope; Fastrach LMA; cervical motion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videolaryngoscope (Active Comparator): Patients intubated with C-Mac D Blade Videolaryngoscope
  Interventions: Device: C-Mac D Blade
- Fastrach LMA (Active Comparator): Patients intubated with Fastrach LMA
  Interventions: Device: Fastrach LMA

INTERVENTIONS:
Device: C-Mac D Blade — Videolaryngoscope
  Arms: Videolaryngoscope
Device: Fastrach LMA — Laryngeal mask airway
  Arms: Fastrach LMA

SUMMARY:
In patients with cervical spine disorders or hernia, in-line stabilization and immobilization during tracheal intubation is used to avoid neck injury. With direct laryngoscopy cranio-cervical motion can result injury. The aim of the study is to compare two different device (C-Mac D blade versus fastrach LMA ) regarding cervical motions during intubation.

DETAILED DESCRIPTION:
In simulated or clinical settings of restricted neck mobility, videolaryngoscopes and fastrach LMA have performed well but neck motion can be occured. Endotracheal intubation will be performed under fluoroscopy. In this study the neck motion angles will be investigated during intubation . The angles will be assessed on fluoroscopy images. A Angle: Angle of the line between occipital protuberance and anterior process of the foramen magnum with the line between central point of spinous process C1 vertebrae and the anterior process of foramen magnum. The reference line for the occiput is defined as a line between the base of the sella and the opisthion (lineA), and the C1 reference line as a line between the lower cortical margin of the spinous process (line B). The C2 reference line is defined as a line between the anterior , inferior margin of the C2 body and the lower cortical margin of the C2 spinous process (lineC). The C5 reference line is a tangent along the superior endplate of the C5 vertebral body (line D). The groups will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of cervical disc herniation ( scheduled cervical discectomy)
2. American Society of Anesthesiology (ASA) physical status I-III patients

Exclusion Criteria:

1. ASA IV patients
2. Age under 18 years, over 70 years
3. Hepatic disease
4. Renal disease
5. Cardiac disease
6. Pregnancy
7. Anticipated difficult airway

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Angle A (degree), Angle B (degree), Angle C(degree) | 30 second
  Angle of the line between occipital protuberance and central point of spinous process of C1 vertebrae. Angle B and Angle C (degree)

CONTACTS AND LOCATIONS:
Overall Officials: derya özkan, assoc prof, Principal Investigator — Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Anesthesiology and Reanimation Clinic Ankara, Turkey Ankara, Turkey
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Ankara, Turkey Ankara, Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozkan D, Altinsoy S, Sayin M, Dolgun H, Ergil J, Donmez A. Comparison of cervical spine motion during intubation with a C-MAC D-Blade(R) and an LMA Fastrach(R). Anaesthesist. 2019 Feb;68(2):90-96. doi: 10.1007/s00101-018-0533-3. Epub 2019 Jan 9. PMID 30627738